CLINICAL TRIAL: NCT00003141
Title: A Pilot Study of Intensive Chemotherapy With Peripheral Stem Cell Support for Infants With Malignant Brain Tumors
Brief Title: Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Infants With Malignant Brain or Spinal Cord Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99703; COG-99703 (Other: Children's Oncology Group); CCG-99703 (Other: Children's Cancer Group); CDR0000065924 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-11-06 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Brain Tumors; Central Nervous System Tumors; Neuroblastoma; Sarcoma
Keywords: childhood infratentorial ependymoma; childhood supratentorial ependymoma; disseminated neuroblastoma; stage 4S neuroblastoma; embryonal childhood rhabdomyosarcoma; childhood high-grade cerebral astrocytoma; childhood choroid plexus tumor; previously untreated childhood rhabdomyosarcoma; untreated childhood brain stem glioma; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood cerebellar astrocytoma; untreated childhood medulloblastoma; newly diagnosed childhood ependymoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma; childhood spinal cord neoplasm; childhood atypical teratoid/rhabdoid tumor; childhood low-grade cerebral astrocytoma; childhood central nervous system choriocarcinoma; childhood central nervous system embryonal tumor; childhood central nervous system germinoma; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Neuroblastoma; Sarcoma; Astrocytoma; Choroid Plexus Neoplasms; Spinal Cord Neoplasms; Rhabdoid Tumor | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; etoposide phosphate; Thiotepa; Vincristine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (combination chemotherapy, PBSC transplant) (Experimental): Pts undergo conventional surgery for diagnosis & max tumor resection. In 6 wks of surgery or when stable pts begin induction chemotherapy(cisplatin IV over 6 hrs on day 0; vincristine sulfate IV on days 0,7,14; cyclophosphamide IV over 1 hr on days 1-2; and etoposide IV over 1 hr on days 0-2. 24 hrs after the last cyclophosphamide dose, pts receive filgrastim (G-CSF) & undergo peripheral blood stem cell harvest 2 days later. Treatment repeats every 21 days for up to 3 crs. Within 6 wks after induction, pts receive consolidation (carboplatin IV over 2 hrs on days 0-1 next esc. doses of thiotepa IV over 2 hrs. Pts undergo peripheral blood stem cell transplantation 48 hrs after last thiotepa dose. Pts receive G-CSF SC daily on days 3-21. Treatment repeats every 21 days for up to 3 crs. Pts with dose-limiting toxicity due to thiotepa are removed from study. Pts are followed at 4 wks, 3 mths for 1 yr, 6 mths for 3 yrs, annually for 3 yrs or until relapse.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide; Drug: thiotepa; Drug: vincristine sulfate; Procedure: conventional surgery; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim — Given IV
  Other Names: GRANULOCYTE COLONY-STIMULATING FACTOR; r-metHuG-CSF; G-CSF
Drug: carboplatin — Given IV
  Other Names: Paraplatin; CBDCA; NSC #241240
Drug: cisplatin — Given IV
  Other Names: Cis-diamminedichloroplatinum II; Platinol-AQ; NSC #119875
Drug: cyclophosphamide — Given IV
  Other Names: CTX; Cytoxan; NSC #026271
Drug: etoposide — Given IV
  Other Names: VP-16; VePesid; Etopophos; NSC #141540
Drug: thiotepa — Given IV
  Other Names: Tespa; Tspa; NSC #639
Drug: vincristine sulfate — Given IV
  Other Names: VCR; Oncovin; NSC #067574
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctors to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy plus peripheral stem cell transplantation in treating infants with malignant brain or spinal cord tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of thiotepa in infants with malignant brain or spinal cord tumors receiving intensive chemotherapy.
* Determine the feasibility and toxicity of intensive chemotherapy with peripheral blood stem cell (PBSC) rescue in these patients.
* Assess the feasibility of harvesting PBSCs in these patients.
* Determine the complete response rate and overall event-free survival rate in patients treated with this regimen.

OUTLINE: This is a pilot, multicenter study.

Patients undergo surgery for diagnosis and maximal tumor resection.

Within 6 weeks of surgery or when stable, patients begin induction chemotherapy comprising cisplatin IV over 6 hours on day 0; vincristine IV on days 0, 7, and 14; cyclophosphamide IV over 1 hour on days 1-2; and etoposide IV over 1 hour on days 0-2. Twenty four hours after the last cyclophosphamide dose, patients receive filgrastim (G-CSF) subcutaneously (SC) and undergo peripheral blood stem cell harvest 2 days later. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Within 6 weeks after induction chemotherapy, patients receive consolidation chemotherapy comprising carboplatin IV over 2 hours on days 0-1 followed immediately by escalating doses of thiotepa IV over 2 hours. Patients then undergo peripheral blood stem cell transplantation 48 hours after the last thiotepa dose. Patients receive G-CSF SC daily on days 3 to 21. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients experiencing dose-limiting toxicity due to thiotepa are removed from the study.

Patients are followed at 4 weeks, every 3 months for 1 year, every 6 months for 3 years, and then annually for 3 years or until relapse.

PROJECTED ACCRUAL: A total of 83 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven malignant brain or spinal cord tumor, including the following:

  * Primitive neuroectodermal tumor
  * Ganglioneuroblastoma
  * Medulloblastoma neuroblastoma
  * Desmoplastic medulloblastoma
  * Medulloepithelioma
  * Ependymoma neuroepithelioma
  * Anaplastic ependymoma germ cell tumor
  * Astrocytoma germinoma
  * Anaplastic astrocytoma
  * Embryonal carcinoma
  * Glioblastoma endodermal sinus tumor
  * Gliosarcoma malignant teratoma
  * Choroid plexus carcinoma
  * Mixed germ cell tumor
  * Cerebellar sarcoma
  * Pineoblastoma
  * Atypical teratoid/rhabdoid tumor
  * Choriocarcinoma
  * Teratoma (malignant or with malignant transformations)
* Diffusely involved brain stem tumors allowed if there is evidence of brain stem glioma by CT scan or MRI

PATIENT CHARACTERISTICS:

Age:

* 6 months to less than 3 years

Performance Status:

* Not specified

Life Expectancy:

* More than 8 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL

Renal:

* Glomerular filtration rate or creatinine clearance greater than 70 mL/min

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior corticosteroids allowed

Radiotherapy:

* No prior radiotherapy

Surgery:

* No more than 6 weeks since prior surgery
* Recovered from prior surgery (stable)

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 1998-03; Primary Completion 2007-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Feasibility | Up to 4 weeks after completion of study treatment
  Demonstrate the feasibility of administering this regimen, to select an acceptable Thiotepa dose for Consolidation therapy, and to document significant toxicities and estimate their overall rates
Maximal tolerated dose of thiotepa for consolidation therapy | 9 weeks
  The dose level will be assigned within 3 working days prior to beginning Consolidation.
Overall rates of significant toxicities including grade IV ototoxicity, electrolytic wasting (grade IV), and hemorrhagic cystitis (grade IV) | Up to 6 years
  Estimates will be obtained using life-table methods with an event defined as the first occurrence of toxicity. Graded using the CCG Toxicity and Complications Criteria.

SECONDARY OUTCOMES:
Event Free Survival | From the time of study entry to the first occurrence of death by any cause, progression or recurrence of disease or occurrence of a second malignant neoplasm, assessed up

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H. Cohen, MD, Study Chair — The Cleveland Clinic
Locations (71):
- United States (66):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics of Minnesota - St. Paul, Saint Paul, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (4):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan